CLINICAL TRIAL: NCT02979418
Title: Pii Ngima: Consequences of Water Insecurity for Maternal and Child Health
Acronym: PEN
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Principal Investigator, Sera Young, Associate Professor, Northwestern University
Other Study IDs: STU00203155
Record Dates: First submitted 2016-11-28; First posted 2016-12-01 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Maternal and Child Health; HIV
Keywords: Water insecurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will implement the validated household-level water insecurity scale developed by study investigators among a cohort of postpartum women in Nyanza, Kenya and will assess a range of outcomes linked to water insecurity, such as viral load, hydration status, maternal depression, stress, food insecurity, and cognitive development.

DETAILED DESCRIPTION:
This study will develop the first well-known household water insecurity scale. Currently, water insecurity cannot be measured at the level of the household or individual, i.e. at the endpoint of water use. Although there are myriad national, regional, community, and hydrological indexes of water availability, to the investigators' knowledge, there is no way of measuring water access at the household or individual levels. Without a comprehensive, validated scale to measure household water insecurity, the scientific, programmatic, and public health communities cannot empirically test the prevalence of household water insecurity access and its potential impacts on economic, nutrition, disease, and psychosocial health pathways and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women >18 years of age with infants enrolled into the Pith Moromo (clinical trials ID: NCT02974972) study
* Infants born to pregnant women enrolled in the cohort study

Exclusion Criteria:

* Individuals <18 years of age that are not infants born to women enrolled in the cohort study

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A cohort of postpartum HIV-infected and -uninfected women (ratio 1:1) who were previously enrolled into the Pith Moromo (clinical trials ID: NCT02974972) research study in Nyanza, Kenya.
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Determine if water insecurity (novel scale) is detrimental to physical health (hemoglobin, hair cortisol, other biomarkers) in ways distinct from food insecurity (Individual Food Insecurity Access Scale) | 2 years
  The investigators are collecting longitudinal cohort data from women who were recruited during pregnancy and have been followed through the first 18 months of the infant's life. Participants are interviewed at regular intervals to gather information on the various pathways through which water insecurity (measured using a novel scale) may be deleterious in ways similar to food insecurity (measured using the Individual Food Insecurity Access Scale).
Determine if water insecurity (novel scale) is detrimental to nutrition (Household Dietary Diversity Scale) in ways distinct from food insecurity (Individual Food Insecurity Access Scale) | 2 years
  The investigators are collecting longitudinal cohort data from women who were recruited during pregnancy and have been followed through the first 18 months of the infant's life. Participants are interviewed at regular intervals to gather information on the various pathways through which water insecurity (measured using a novel scale) may be deleterious in ways similar to food insecurity (measured using the Individual Food Insecurity Access Scale).
Determine if water insecurity (novel scale) is detrimental to psychosocial health (Perceived Stress Scale, Center for Epidemiology Depression (CES-D) scale, etc.), in ways distinct from food insecurity (Individual Food Insecurity Access Scale) | 2 years
  The investigators are collecting longitudinal cohort data from women who were recruited during pregnancy and have been followed through the first 18 months of the infant's life. Participants are interviewed at regular intervals to gather information on the various pathways through which water insecurity (measured using a novel scale) may be deleterious in ways similar to food insecurity (measured using the Individual Food Insecurity Access Scale).
Determine if water insecurity (novel scale) is detrimental to economic security (asset index) in ways distinct from food insecurity (Individual Food Insecurity Access Scale) | 2 years
  The investigators are collecting longitudinal cohort data from women who were recruited during pregnancy and have been followed through the first 18 months of the infant's life. Participants are interviewed at regular intervals to gather information on the various pathways through which water insecurity (measured using a novel scale) may be deleterious in ways similar to food insecurity (measured using the Individual Food Insecurity Access Scale).

SECONDARY OUTCOMES:
Determining if water insecurity (measured using a novel tool) will differ by HIV status | 2 years
  The investigators collected longitudinal data to assess water insecurity among the cohort (using a novel tool) and will compare the prevalences and impacts of water insecurity by HIV status

REFERENCES:
- [Result] Krumdieck NR, Collins SM, Wekesa P, Mbullo P, Boateng GO, Onono M, Young SL. Household water insecurity is associated with a range of negative consequences among pregnant Kenyan women of mixed HIV status. J Water Health. 2016 Dec;14(6):1028-1031. doi: 10.2166/wh.2016.079. PMID 27959881
- [Result] Brooks YM, Collins SM, Mbullo P, Boateng GO, Young SL, Richardson RE. Evaluating Human Sensory Perceptions and the Compartment Bag Test Assays as Proxies for the Presence and Concentration of Escherichia coli in Drinking Water in Western Kenya. Am J Trop Med Hyg. 2017 Oct;97(4):1005-1008. doi: 10.4269/ajtmh.16-0878. Epub 2017 Jul 27. PMID 28749760
- [Result] Miller JD, Fitzgerald KG, Smith AL, Young SL. Geophagy among a Cohort of Kenyan Women with Mixed HIV Status: A Longitudinal Analysis. Am J Trop Med Hyg. 2019 Sep;101(3):654-660. doi: 10.4269/ajtmh.19-0149. PMID 31333167
- [Result] Boateng GO, Workman CL, Miller JD, Onono M, Neilands TB, Young SL. The syndemic effects of food insecurity, water insecurity, and HIV on depressive symptomatology among Kenyan women. Soc Sci Med. 2022 Feb;295:113043. doi: 10.1016/j.socscimed.2020.113043. Epub 2020 May 15. PMID 32482382
- [Result] Collins SM, Mbullo Owuor P, Miller JD, Boateng GO, Wekesa P, Onono M, Young SL. 'I know how stressful it is to lack water!' Exploring the lived experiences of household water insecurity among pregnant and postpartum women in western Kenya. Glob Public Health. 2019 May;14(5):649-662. doi: 10.1080/17441692.2018.1521861. Epub 2018 Sep 20. PMID 30231793
- [Derived] Alvarez GG, Miller JD, Santoso MV, Wekesa P, Owuor PM, Onono M, Young SL. Prevalence and Covariates of Food Insecurity Across the First 1000 Days Among Women of Mixed HIV Status in Western Kenya: A Longitudinal Perspective. Food Nutr Bull. 2021 Sep;42(3):319-333. doi: 10.1177/0379572121999024. Epub 2021 May 20. PMID 34011176
- [Derived] Benzaken CL, Miller JD, Onono M, Young SL. Development of a cumulative metric of vaccination adherence behavior and its application among a cohort of 12-month-olds in western Kenya. Vaccine. 2020 Apr 16;38(18):3429-3435. doi: 10.1016/j.vaccine.2020.03.011. Epub 2020 Mar 14. PMID 32184035